CLINICAL TRIAL: NCT01840501
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single- and Multiple-Doses of JNJ-42721458 in Healthy Male Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-42721458 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR101337; 42721458EDI1001 (Other: Janssen Research & Development, LLC); 2013-000557-47 (EudraCT Number)
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Healthy; JNJ-42721458; Male; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; Immunogenicity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (18):
- Part 1: Panel 1 (0.1 mg JNJ-42721458) (Experimental): 6 participants will receive a single dose of 0.1 mg of JNJ-42721458.
  Interventions: Drug: JNJ-42721458 (single dose)
- Part 1: Panel 2 (0.3 mg JNJ-42721458) (Experimental): 6 participants will receive a single dose of 0.3 mg of JNJ-42721458.
  Interventions: Drug: JNJ-42721458 (single dose)
- Part 1: Panel 3 (1.0 mg JNJ-42721458) (Experimental): 6 participants will receive a single dose of 1.0 mg of JNJ-42721458.
  Interventions: Drug: JNJ-42721458 (single dose)
- Part 1: Panel 4 (2.5 mg JNJ-42721458) (Experimental): 6 participants will receive a single dose of 2.5 mg of JNJ-42721458.
  Interventions: Drug: JNJ-42721458 (single dose)
- Part 1: Panel 5 (5.0 mg JNJ-42721458) (Experimental): 6 participants will receive a single dose of 5.0 mg of JNJ-42721458.
  Interventions: Drug: JNJ-42721458 (single dose)
- Part 1: Panel 6 (10.0 mg JNJ-42721458) (Experimental): 6 participants will receive a single dose of 10.0 mg of JNJ-42721458.
  Interventions: Drug: JNJ-42721458 (single dose)
- Part 1: Panel 7 (20.0 mg JNJ-42721458) (Experimental): 6 participants will receive a single dose of 20.0 mg of JNJ-42721458.
  Interventions: Drug: JNJ-42721458 (single dose)
- Part 1: Panel 8 (Experimental): 6 participants will receive a single dose JNJ-42721458, the dose will be determined after completion of panels 1-7 in Part 1.
  Interventions: Drug: JNJ-42721458 (single dose)
- Part 1: Panel 9 (Experimental): 6 participants will receive a single dose JNJ-42721458, the dose will be determined after completion of panels 1-8 in Part 1.
  Interventions: Drug: JNJ-42721458 (single dose)
- Part 1: Panel 10 (Experimental): 6 participants will receive a single dose JNJ-42721458, the dose will be determined after completion of panels 1-9 in Part 1.
  Interventions: Drug: JNJ-42721458 (single dose)
- Part 1: Placebo (Placebo Comparator): 2 participants from each panel will receive a single dose of placebo.
  Interventions: Drug: Placebo (single dose)
- Part 2: Panel 1 (5.0 mg JNJ-42721458) (Experimental): 6 participants will receive multiple doses of 5.0 mg of JNJ-42721458.
  Interventions: Drug: JNJ-42721458 (multiple doses)
- Part 2: Panel 2 (10.0 mg JNJ-42721458) (Experimental): 6 participants will receive multiple doses of 10.0 mg of JNJ-42721458.
  Interventions: Drug: JNJ-42721458 (multiple doses)
- Part 2: Panel 3 (Experimental): 6 participants will receive multiple doses of JNJ-42721458, the dose will be determined after completion of panels 1-2 in Part 2.
  Interventions: Drug: JNJ-42721458 (multiple doses)
- Part 2: Panel 4 (Experimental): 6 participants will receive multiple doses of JNJ-42721458, the dose will be determined after completion of panels 1-3 in Part 2.
  Interventions: Drug: JNJ-42721458 (multiple doses)
- Part 2: Panel 5 (Experimental): 6 participants will receive multiple doses of JNJ-42721458, the dose will be determined after completion of panels 1-4 in Part 2.
  Interventions: Drug: JNJ-42721458 (multiple doses)
- Part 2: Panel 6 (Experimental): 6 participants will receive multiple doses of JNJ-42721458, the dose will be determined after completion of panels 1-5 in Part 2.
  Interventions: Drug: JNJ-42721458 (multiple doses)
- Part 2: Placebo (Placebo Comparator): 2 participants from each panel will receive multiple doses of placebo.
  Interventions: Drug: Placebo (multiple doses)

INTERVENTIONS:
Drug: JNJ-42721458 (single dose) — JNJ-42721458 will be administered subcutaneously (an injection under the skin) as single doses, starting from 0.1 mg.
  Arms: Part 1: Panel 1 (0.1 mg JNJ-42721458); Part 1: Panel 10; Part 1: Panel 2 (0.3 mg JNJ-42721458); Part 1: Panel 3 (1.0 mg JNJ-42721458); Part 1: Panel 4 (2.5 mg JNJ-42721458); Part 1: Panel 5 (5.0 mg JNJ-42721458); Part 1: Panel 6 (10.0 mg JNJ-42721458); Part 1: Panel 7 (20.0 mg JNJ-42721458); Part 1: Panel 8; Part 1: Panel 9
Drug: JNJ-42721458 (multiple doses) — JNJ-42721458 will be administered subcutaneously (an injection under the skin) once daily, starting with a dose of 5.0 mg.
  Arms: Part 2: Panel 1 (5.0 mg JNJ-42721458); Part 2: Panel 2 (10.0 mg JNJ-42721458); Part 2: Panel 3; Part 2: Panel 4; Part 2: Panel 5; Part 2: Panel 6
Drug: Placebo (single dose) — Matching placebo will be administered subcutaneously (an injection under the skin) as a single dose in Part 1.
  Arms: Part 1: Placebo
Drug: Placebo (multiple doses) — Matching placebo will be administered subcutaneously (an injection under the skin) once daily for 10 days in Part 2.
  Arms: Part 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (what the body does to the medication), potential immunogenicity (ability to induce an immune response), and pharmacodynamics (what the drug does to the body) after administration of JNJ-42721458 in healthy adult male participants.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), double-blind (neither physician nor participant knows the identity of the assigned treatment), placebo-controlled (an inactive substance that is compared with a medication to test whether the medication has a real effect in a clinical study), single-ascending (increasing) dose and multiple-ascending dose study of JNJ-42721458 compound in healthy males. The study is divided in two parts. Part 1 is a single-ascending dose (SAD) study which will include up to 10 panels (using ascending doses starting from 0.1 mg) in which a single dose of the study medication will be administered on Day 1. Part 2 is a multiple-ascending dose (MAD) study which will include approximately 6 panels (using ascending doses starting from 5.0 mg) in which multiple doses of study medication will be administered once daily for 10 days.

Part 2 will be initiated after completion of dosing and all relevant evaluations from Part 1. In each panel of Part 1 and 2, 6 participants will be randomly assigned to receive JNJ-42721458 and 2 participants randomly assigned to placebo. Safety evaluations will include assessment of adverse events, physical examinations, laboratory tests, vital signs, electrocardiograms, cardiac telemetry and evaluation of injection sites which will be monitored throughout the study. The total study duration for each participant will be approximately 6-7 weeks in Part 1 and 7-8 weeks for each participant in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (weight kg/m2) between 18 and 30 kg/m2, and body weight not less than 50 kg
* Participant is judged to be generally in good health based on medical history, physical examination, vital signs and laboratory safety tests
* Blood pressure between 90 and 135 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic
* A 12-lead electrocardiogram consistent with normal cardiac conduction and function

Exclusion Criteria:

* History of or current clinically significant medical illness
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or on Day -1 (at admission to the study center)
* Estimated creatinine clearance of less than or equal to 80 mL/min
* Clinically significant abnormal physical examination, vital signs or 12 lead electrocardiogram at screening or on Day -1
* Participant demonstrates orthostatic change in vital signs measurements on screening or predose while going from a semi recumbent to standing position
* History of significant multiple and/or severe allergies (including latex allergies) or known history of clinically significant allergies to polyethylene glycol (PEG) containing or other PEGylated products

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Part 1 and 2: Number of participants with adverse events | Up to 17 weeks
  Number of participants with adverse events will be used as a measure of safety and tolerability.
Part 1 and 2: Maximum observed concentration (Cmax) of JNJ-42721458 | Up to Day 10 (for Part 1) and Day 27 (for Part 2)
Part 1 and 2: Time to reach the maximum plasma concentration (tmax) of JNJ-42721458 | Up to Day 10 (for Part 1) and Day 27 (for Part 2)
Part 1 and 2: Area under the concentration-time curve of JNJ-42721458, from time 0 to infinity, with extrapolation of the terminal phase | Up to Day 10 (for Part 1) and Day 27 (for Part 2)
Part 1 and 2: Area under the concentration-time curve of JNJ-42721458 during a dosing interval at steady state | Up to Day 10 (for Part 1) and Day 27 (for Part 2)
Part 1 and 2: Terminal half-life (t1/2) of JNJ-42721458 | Up to Day 10 (for Part 1) and Day 27 (for Part 2)
Part 1 and 2: Apparent systemic clearance of drug after subcutaneous administration of JNJ-42721458 | Up to Day 10 (for Part 1) and Day 27 (for Part 2)
Part 1 and 2: Apparent volume of distribution after subcutaneous administration of JNJ-42721458 | Up to Day 10 (for Part 1) and Day 27 (for Part 2)
Part 1 and 2: Plasma levels of antibodies to JNJ-42721458 for evaluation of potential immunogenicity | Up to Day 10 (for Part 1) and Day 27 (for Part 2)

SECONDARY OUTCOMES:
Part 1 and 2: Change from baseline in resting heart rate | Up to Day 10 (for Part 1) and Day 27 (for Part 2)
Part 1 and 2: Change from baseline in resting peripheral blood pressure | Up to Day 10 (for Part 1) and Day 27 (for Part 2)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium